CLINICAL TRIAL: NCT05257460
Title: Closing the Loop in Adults With Type 1 Diabetes Under Free Living Conditions. A Double-blinded, Single Centre, Randomised, Two-period, Crossover Extension Phase to Evaluate Home Use of Closed-loop Applying Ultra-rapid Insulin Lispro Versus Standard Insulin Lispro (Phase 4).
Brief Title: Closing the Loop in Adults With Type 1 Diabetes Under Free Living Conditions (AP@Home04_Phase 4)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor of Metabolic Technology, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 136248_Version_7.1
Record Dates: First submitted 2022-02-07; First posted 2022-02-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop using standard rapid-acting insulin lispro (Active Comparator): Unsupervised home use of day and night hybrid closed loop insulin delivery system (CamAPS FX) for 8 weeks using standard rapid-acting insulin lispro.
  The CamAPS FX closed-loop system comprises Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA), an Android smartphone hosting CamAPS FX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system.
  Interventions: Device: Hybrid closed-loop using standard insulin lispro
- Closed-loop using ultra-rapid insulin lispro (Experimental): Unsupervised home use of day and night hybrid closed loop insulin delivery system (CamAPS FX) for 8 weeks using ultra-rapid insulin lispro.
  The CamAPS FX closed-loop system comprises Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA), an Android smartphone hosting CamAPS FX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system.
  Interventions: Device: Hybrid closed-loop using ultra-rapid insulin lispro

INTERVENTIONS:
Device: Hybrid closed-loop using ultra-rapid insulin lispro — Hybrid closed-loop using ultra-rapid insulin lispro
  Arms: Closed-loop using ultra-rapid insulin lispro
Device: Hybrid closed-loop using standard insulin lispro — Hybrid closed-loop using standard insulin lispro
  Arms: Closed-loop using standard rapid-acting insulin lispro

SUMMARY:
The main objective of this study is to determine whether home use of day and night closed loop insulin delivery under free living conditions applying ultra-rapid insulin lispro (Lyumjev) is superior to home use of closed-loop applying standard insulin lispro (Humalog).

This is a double-blind, single-centre, randomised, crossover design study, involving a run-in period followed by two study periods during which glucose levels will be controlled either by an automated closed-loop system using standard rapid acting Humalog or by an automated closed-loop system using ultra-rapid Lispro in random order.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. Subjects will have regular contact with the study team during the home study phase including 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM during home stay. Secondary outcomes include time spent with glucose levels above and below target, as recorded by CGM, and other CGM based metrics.

DETAILED DESCRIPTION:
Purpose of clinical trial The purpose is to determine whether home use of day and night closed loop applying ultra-rapid insulin lispro is superior to home use of closed loop applying standard insulin lispro.

Study objectives The study objective is to compare day and night automated closed-loop glucose control using ultra-rapid insulin lispro with closed loop control using standard insulin lispro.

EFFICACY: The objective is to assess the efficacy of day and night automated closed-loop glucose control applying standard insulin lispro in maintaining CGM glucose levels within the target range from 3.9 to 10.0 mmol/l, as compared to day and night closed-loop using ultra-rapid acting insulin lispro.

SAFETY: The objective is to evaluate the safety of day and night automated closed-loop glucose control in terms of episodes of severe hypoglycaemia, hyperglycaemia and other adverse events and adverse device effects.

UTILITY: The objective is to determine the percentage of time when closed-loop was operational, and usability and acceptance of the closed-loop system.

Study Design A double-blind, single-centre, randomised, two-period crossover study, contrasting day and night automated closed-loop glucose control applying standard insulin lispro with day and night closed-loop control applying ultra-rapid acting insulin lispro.

Study Efficacy Endpoints The primary outcome is the time spent in the target glucose range from 3.9 to 10.0 mmol/l based on CGM glucose levels during the free living phase.

Secondary outcomes include time spent above and below the target glucose range, based on CGM levels.

Safety Evaluation Frequency of severe hypoglycaemic episodes as defined by American Diabetes Association, frequency of severe hyperglycaemia (>20 mmol/L) and / or significant ketosis (plasma ketones >3mmol/l) and nature and severity of other adverse events.

Utility Evaluation Percentage of time spent in closed-loop. Usability and acceptance of the closed-loop system will be assessed using a patient experience questionnaire at the end of the second intervention. Additionally, human factor questionnaires will be administered following recruitment and at the end of each intervention arm.

Sample Size 24 adults completing the study. Up to 30 subjects will be recruited to allow for dropouts.

Maximum duration of study for a subject 20 weeks (5 months)

Recruitment The subjects will be recruited through the adult diabetes outpatient clinics or other established methods at the participating centre.

Consent Participants will be asked to provide written informed consent.

Baseline Assessment Eligible subjects will undergo a baseline evaluation including a blood sample for the measurement of HbA1c, renal, liver function, full blood count, thyroid function and coeliac antibody screen (if not done in the previous 3 months). Urine pregnancy test will be done in females. Human factor questionnaires will be administered.

Study Training and Run-in Period Training sessions on the use of study CGM, insulin pump and closed-loop system will be provided by the research team. During the 2-4 weeks run-in period, subjects will use study CGM and insulin pump and will have regular contact with the research team. At the end of the run-in period, for compliance and to assess the ability of the subject to use the CGM and study pump safely, before the start of the first home study phase, at least 7 days of CGM data need to be recorded and safe use of study insulin pump demonstrated. CGM and insulin pump data during the run-in period will be used to assess baseline glucose control and optimise treatment before the start of the first home study phase.

Competency Assessment Competency on the use of study insulin pump, study CGM and closed-loop system will be evaluated using a competency assessment tool developed by the research team. Further training may be delivered as required.

Randomisation Eligible subjects will be randomised using randomisation software to the initial use of closed-loop with ultra-rapid insulin lispro followed by closed-loop with standard insulin lispro or the alternate order.

Automated closed-loop Training on the use of closed-loop will be provided by the research team. Automated closed-loop control will be commenced and during the training; the participant will operate the system under the supervision of the clinical team. Competency on the use of closed-loop system will be evaluated. Subjects will be advised to use automated closed-loop system for next 8 weeks

Cross-over Assessment At the end of the first intervention human factor questionnaires will be administered.

There will be no washout period in phase 4 extension.

End of study assessments A patient experience questionnaire will be given at the end of the second intervention. Additionally human factor questionnaires will be administered.

Procedures for safety monitoring during trial Standard operating procedures for monitoring and reporting of all adverse events and adverse device events will be in place, including serious adverse events (SAE), serious adverse device effects (SADE) and specific adverse events (AE) such as severe hypoglycaemia.

Criteria for withdrawal of patients on safety grounds

A subject may terminate participation in the study at any time without necessarily giving a reason and without any personal disadvantage. An investigator can stop the participation of a subject after consideration of the benefit/risk ratio. Possible reasons are:

Serious adverse events Significant protocol violation or noncompliance Failure to satisfy competency assessment Decision by the investigator, or the sponsor, that termination is in the subject's best medical interest Pregnancy, planned pregnancy, or breast feeding Allergic reaction to insulin Technical grounds (e.g. subject relocates)

ELIGIBILITY:
Inclusion Criteria:

* The subject has type 1 diabetes as defined by WHO
* The subject is 18 years of age or older
* The subject will have been on an insulin pump for at least 6 months with good knowledge of insulin self-adjustment including carbohydrate counting
* The subject is treated with one of the rapid acting or ultra-rapid acting insulin analogues (Insulin Aspart, faster acting insulin Aspart, Insulin Lispro or Insulin Glulisine)
* HbA1c <10% (86mmol/mol) based on analysis from central laboratory or equivalent
* The subject is willing to wear closed-loop system at home and at work place
* The subject is willing to follow study specific instructions including the use of bolus calculator for all meals / snacks
* The subject is willing to upload pump and CGM data at regular intervals
* Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening.

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
* Known or suspected allergy against insulin or previous reaction to FiAsp
* More than one episode of severe hypoglycaemia as defined by American Diabetes Association (42) in preceding 12 months (Severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions including episodes of hypoglycaemia severe enough to cause unconsciousness, seizures or attendance at hospital.)
* Total daily insulin dose > 2 IU/kg/day
* Subject is pregnant or breast feeding or planning pregnancy within next 10 months
* Severe visual impairment
* Severe hearing impairment
* Lack of reliable telephone facility for contact
* Subject not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on continuous glucose monitoring (CGM) | 8-weeks

SECONDARY OUTCOMES:
Time spent above target glucose range (>10.0 mmol/l) based on continuous glucose monitoring (CGM) | 8-weeks
Time spent below target glucose range (<3.9 mmol/l) based on continuous glucose monitoring (CGM) | 8-weeks
Average of glucose levels based on continuous glucose monitoring | 8-weeks
Standard deviation of glucose levels based on continuous glucose monitoring | 8-weeks
Coefficient of variation of glucose levels based on continuous glucose monitoring | 8-weeks
The time with glucose levels <3.0mmol/l based on continuous glucose monitoring | 8-weeks
The time with glucose levels in significant hyperglycaemia, as based on continuous glucose monitoring (glucose levels >16.7 mmol/l) | 8-weeks
Total daily insulin dose (units/day) | 8-weeks
Total basal insulin dose (units/day) | 8-weeks
Total bolus insulin dose (units/day) | 8-weeks

OTHER OUTCOMES:
Safety evaluation will comprise the number of episodes of hypoglycaemia, significant ketonemia (>3.0mmol/l) as well as nature and severity of any other adverse events. | Through study completion (up to 5 months)
Utility evaluation is the frequency and duration of use of the closed-loop system at home | 8-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to rh347@cam.ac.uk and may be submitted up to 36 months following article publication.

REFERENCES:
- [Derived] Haliloglu B, Boughton CK, Lakshman R, Ware J, Nwokolo M, Thabit H, Mader JK, Bally L, Leelarathna L, Wilinska ME, Allen JM, Hartnell S, Evans ML, Hovorka R. Postprandial Glucose Excursions with Ultra-Rapid Insulin Analogs in Hybrid Closed-Loop Therapy for Adults with Type 1 Diabetes. Diabetes Technol Ther. 2024 Jul;26(7):449-456. doi: 10.1089/dia.2023.0509. Epub 2024 Feb 27. PMID 38315506
- [Derived] Nwokolo M, Lakshman R, Hartnell S, Alwan H, Ware J, Allen JM, Wilinska ME, Evans ML, Hovorka R, Boughton CK. CamAPS FX Hybrid Closed-Loop with Ultra-Rapid Lispro Compared with Standard Lispro in Adults with Type 1 Diabetes: A Double-Blind, Randomized, Crossover Study. Diabetes Technol Ther. 2023 Dec;25(12):856-863. doi: 10.1089/dia.2023.0262. PMID 37823892